CLINICAL TRIAL: NCT00513032
Title: Effects of Methylene Blue on Propofol Requirement During Anaesthesia Induction and Surgery
Brief Title: Interaction Between Anaesthetics and Methylene Blue
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Other Study IDs: 02-081(02-006)
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2007-08-08 (Estimated); Status verified 2007-08

CONDITIONS: Hyperparathyroidism
Keywords: propofol; anaesthesia induction; parathyroidectomy; methylene blue; General anesthesia
MeSH Terms: conditions — Hyperparathyroidism | interventions — Methylene Blue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- methylene blue
  Interventions: Drug: methylene blue
- C
  Interventions: Drug: methylene blue

INTERVENTIONS:
Drug: methylene blue — 5mg.kg-1 methylene blue in 250 ml 5% glucose-saline, administered intravenously approximately 60 min before anaesthesia induction

SUMMARY:
We hypothesized that pre-treatment with methylene blue could potentiate the effects of general anaesthetic agents in patients undergoing parathyroidectomy

DETAILED DESCRIPTION:
Sample and study design The local ethics committee granted approval for this study and informed written consent will be obtained from all participants. We will study ASA grade I or II patients, aged between 45 and 73 years who were free from cardiovascular and pulmonary diseases. Patients with psychiatric disorders or drug abuse as well as those weighing 20% more or less than their ideal body weight will all be excluded.

The interventional group will consist of 11 patients scheduled for elective parathyroidectomy who will receive MB infusion (5mg.kg-1 in 250 ml 5% glucose-saline) approximately 60 min before anaesthesia induction. A further 11 patients scheduled for unilateral thyroid lobectomy without MB pre-treatment will be recruited as controls. They will present with normal thyroid tests and will carefully be selected in an attempt to match the intervention group on the basis of age, weight and sex. Both types of surgical procedures will be performed by the same surgical team.

Anaesthesia and surgery All patients will be premedicated with oral midazolam 7.5 mg and they will receive a loading dose of lactate-ringer solution (5 ml.kg-1) intravenously after arrival in the operating theatre. The standard anaesthetic monitoring will comprise non-invasive blood pressure, ECG, pulsed oxygen saturation and end-tidal carbon dioxide. Processed EEG parameters will be acquired with a BIS monitor, using surface electrodes, with impedance maintained at less than 5kΩ to ensure adequate signal quality. Raw EEG data from two channels (F7-CZ and F8-CZ) will be processed by company proprietary software and the BIS values (calculated for each 4-sec epoch) will be continuously displayed along with the trend line.

Propofol will be infused using a commercially available TCI system loaded with Schneider's 3-compartment pharmacokinetic model wherein the individual patient's age, height and weight will be programmed. The target effect-site concentration of propofol will be computed to yield a time to peak effect of 1.6 min, which has been confirmed clinically.

During anaesthesia induction, the patients will breath an air-oxygen mixture through a face mask. The target effect-site concentration of propofol will first be set at 0.5 ng.ml-1 and it will be increased by 0.2 ng.ml-1 every 2 min until the clinical endpoint will be achieved (loss of consciousness and unresponsiveness). Then, ventilation will be assisted manually and the trachea will be intubated after the intravenous administration of fentanyl (100 mcg) and rocuronium (0.7 mg.kg-1).

During anaesthesia maintenance, the effect-site concentration of propofol will be targeted to achieve BIS values between 30 and 60. Additional fentanyl, rocuronium or vasopressor agents (ephedrine) will be given at the discretion of the attending anaesthetist.

Measurements When each patient will be comfortable on the operating table, baseline measurements of BIS, mean arterial pressure (MAP), heart rate (HR) and pulsed oxygen saturation (SpO2) will be taken.

During propofol induction, BIS values, MAP, HR and SpO2 will be recorded every 1-min and the Observer's Assessment of Alertness/Sedation (OAAS) rating scale will be recorded after each equilibration period (score 5=awake and responds readily to name spoken in normal tone; 4= lethargic response to name in normal tone; 3=response only after name is called loudly and/or repeatedly; 2= response only after name is called loudly and after mild shaking; 1= dose not respond when name is called and after mild shaking).

During surgery and anaesthesia maintenance, BIS values and the effect-site concentration of propofol will be recorded each 5-min.

Other recorded data will include the doses of propofol required for anaesthesia induction and maintenance, the total amount of vasopressor and the time until anaesthesia emergence and readiness for tracheal extubation.

Statistics Assuming that MB pre-treatment would reduce the requirement of propofol by 25%, power analysis with alpha = 0.05, beta = 0.8, shows that we would need to study at least 10 patients in each group. The computer program SAS 8.0 for Windows will be used for all data analyses. Parametric data will be analysed by two-way ANOVA. Unpaired Student t-tests, Chi-squared tests and Fisher's exact probability tests will be used as appropriate for comparison between groups. All values are expressed as mean (M), standard deviation (SD) and statistical significance will be accepted at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing parathyroidectomy or partial thyroidectomy

Exclusion Criteria:

* Psychiatric disorders
* Drug abuse
* Weight 20% more or less than ideal body weight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-01; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Licker, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Service d'Anesthésiologie, Hôpitaux Universitaires de Genève, Rue Micheli-du-Crest, Geneva, Switzerland